CLINICAL TRIAL: NCT05873140
Title: Healthy Thai Project With Bangkoknoi Model: Fatless Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Phunchai Charatcharoenwitthaya, Professor, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Si 1000/2021
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Continuously receiving education (video clips and infographics) via application LINE
  Interventions: Behavioral: application LINE
- Control group (No Intervention): No application LINE

INTERVENTIONS:
Behavioral: application LINE — Online lifestyle modification education for weight loss
  Arms: Study group

SUMMARY:
The goal of this interventional study is to make people in a community realize negative effects of obesity on health, and how to tackle it by adopting a lifestyle modification for weight reduction. Adults aged 20 years old or more with obesity (BMI ≥ 25 kg/m2) or waist circumference ≥ 80 cm in women and ≥ 90 cm in men were recruited. All participants received an educational session of lifestyle modification for weight reduction on the first day of study. Participants were then assigned to either continuously receive education (video clips and infographics) via application LINE, or no further education. The main questions it aims to answer are:

1. Whether or not an educational session of lifestyle modification leads to weight reduction.
2. Whether or not a weight loss by a continuous education via an online application is more effective than not receiving it.

ELIGIBILITY:
Inclusion Criteria:

* Obesity (BMI ≥ 25 kg/m2)
* Waist circumference ≥ 80 cm in women and ≥ 90 cm in men

Exclusion Criteria:

* Contraindications for bioelectrical impedance analysis
* Active cancer
* No available health data

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-06-26 (Actual); Primary Completion 2023-04-02 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
Body weight change | 6 months after intervention
  Body weight change

CONTACTS AND LOCATIONS:
Overall Officials: Phunchai Charatcharoenwitthaya, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand